CLINICAL TRIAL: NCT01915979
Title: Role of Biological Therapy in Rotator Cuff Tendinopathy. Effectiveness of Plasma Rich in Growth Factors Regarding Functional Capacity and Pain Compared With the Conventional Treatment Using Steroids
Brief Title: Effect of Plasma Rich in Growth Factors in Rotator Cuff Tendinopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Principe de Asturias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUPA-EC-02-2012; 2012-001056-19 (EudraCT Number)
Record Dates: First submitted 2013-07-18; First posted 2013-08-05 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: plasma rich in growth factors, tendinopathy, traumatology; ,rotator cuff, effectiveness, plasma rich in platelets
MeSH Terms: conditions — Tendinopathy | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plasma rich in growth factors (PRGF) (Experimental): This group will receive a total of three intraarticular injections of 6-8 ml. One injection every two weeks.
  Interventions: Biological: Plasma rich in growth factors (PRGF)
- Celestone cronodose (bethametasone) (Active Comparator): This group will receive a total of three intraarticular injections of 2ml. One injection every two weeks.
  Interventions: Drug: Celestone cronodose (Bethametasone)

INTERVENTIONS:
Biological: Plasma rich in growth factors (PRGF)
  Arms: Plasma rich in growth factors (PRGF)
Drug: Celestone cronodose (Bethametasone)
  Arms: Celestone cronodose (bethametasone)

SUMMARY:
The overall objective of the study is to assess the effectiveness of the treatment of degenerative rotator cuff tendinopathy using the application of plasma rich in growth factors (PRGF).

Main objective:

To show more effectiveness after 6 months of treatment with PRGF, with an improvement in the reference test of more than 15% compared to the treatment with corticosteroids.

Secondary objective:

* To assess the efficacy of the treatment after 12 months.
* Quantification of platelet levels in patients treated with plasma rich in growth factors and its correlation with the clinical effect.

DETAILED DESCRIPTION:
Study Group. PRGF

Blood extraction was performed in the pre-surgical area using a vacuum system. A total of 20 ml of blood (4 samples of 5 ml) per patient was collected in sterile sodium citrate tubes. PRGF was obtained following Anitua's technique. The tubes with citrated blood were centrifuged at 1,800 rpm for 8 min to obtain a concentrate of platelets suspended in plasma, which was separated into three fractions. Pipetting was carried out with extreme care in all steps, particularly in the last fraction where, in order to avoid inflammation, leukocytes present in the lowermost portion of the centrifuged plasma were not aspirated. PRGF was activated by adding calcium chloride 10%,immediately before infiltration. The proportion required for PRGF activation is 50 ml of activator per 1,000 ml of PRGF. Separation of plasma into three fractions and subsequent activation of the fractions for injection was performed in a laminar flow chamber.

Between the collection of blood and its subacromial administration must not exceed 90 minutes to avoid contamination.

Control group: Celestone Cronodose® (bethametasone).

They were given 3 infiltrations of 2 cc of Celestone cronodose® (bethametasone) every 21 days (If necessary, it could be administered after an application of a small quantity of a local anaesthetic).

ELIGIBILITY:
Inclusion Criteria:

* Patients within 40 -70 years old.
* Both sex
* Moderate to severe symptoms according to the QuickDASH scale during the last 3 months.
* Patients with tendinitis, inflammatory or calcium, tendinosis or partial tears of the rotator cuff, diagnosed by ultrasound or MRI, evaluated by an expert radiologist and independent of research team.
* Patients resistant to conservative treatment.

Exclusion Criteria:

* Patients with complete tear of the rotator cuff diagnosed by ultrasound or MRI.
* Patients who have previously received treatment with infiltrations in the last 6 months.
* Patients with poorly controlled arterial Hypertension (AHT) and Diabetes mellitus.
* Allergic to some of the components of Celestone Cronodose ®, either the drug or some of the excipients.
* Patients on anticoagulants or antiplatelet therapy which cannot be reversed temporarily for the infiltrations.
* Positive serology for sifilis, hepatitis B, hepatitis C or IHV I/II.
* Uncapable to understand health questionnaires and / or complete them properly.
* Women who might be pregnant and don't have a negative pregnancy test at the start of the study.
* Breastfeeding women.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
15% of change in the score of the UCLA scale | Baseline and 6 months
15% of change in the score of the QuickDash scale | Baseline and 6 months

SECONDARY OUTCOMES:
changes in the UCLA, Quickdash and Constant scales | 12 months
Concentration of the platelet levels in the plasma administered and its relationship with the clinical effect measured with the UCLA and QuickDash scales. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Victor Vaquerizo, MD, PhD, Principal Investigator — Hospital Universitario Principe de Asturias
Locations (1):
- Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid, Spain